CLINICAL TRIAL: NCT02798016
Title: Treatment of Atrophic Acne Scars With Platelet-Rich Plasma Alone or in Combination With Skin Needling: A Randomized Controlled Trial
Brief Title: Treatment of Atrophic Acne Scars With Platelet-Rich Plasma and Skin Needling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDMS-Dermat-01-2016
Record Dates: First submitted 2016-05-13; First posted 2016-06-14 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Atrophic Acne Scars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet-Rich Plasma alone (Experimental): The scars will be injected with Platelet-Rich Plasma alone.
  Interventions: Procedure: Platelet-Rich Plasma
- Platelet-Rich Plasma with micro-needling (Active Comparator): The scars will be dealt with using micro-needling as well as injecting Platelet-Rich Plasma
  Interventions: Procedure: Platelet-Rich Plasma; Procedure: Micro-needling

INTERVENTIONS:
Procedure: Platelet-Rich Plasma — This Platelet-Rich Plasma will be taken from each patient and is going to be used in the treatment of atrophic acne scars
Procedure: Micro-needling — Micro-needling will be applied on the acne scars in one side of the face.
  Arms: Platelet-Rich Plasma with micro-needling

SUMMARY:
Investigators will collect blood specimens from the participating patients and then blood samples will be centrifuged in order to collect platelet-rich plasma which is going to be injected in the atrophic acne scars. A split-face design is going to used in this randomized controlled trial. In the control side of the face, micro-needling to the skin will occur using a specific tool (Dermapen).

DETAILED DESCRIPTION:
Atrophic acne scar is a common problem with a challenging treatment. Platelet-rich plasma (PRP) is an autologous preparation of platelets in concentrated plasma that may be beneficial in the treatment of atrophic acne scars by promoting collagen deposition.

Skin needling is a technique that uses a sterile micro needles to puncture the skin and release growth factors. The combination of skin needling and PRP could enhance the efficacy of both modalities.

ELIGIBILITY:
Inclusion Criteria:

* Atrophic acne scars on both sides of the face

Exclusion Criteria:

* patients with active acne, herpes labialis, or bacterial infection; warts on the face, actinic keratosis, or skin cancer
* systemic retinoids intake in the previous 6 months,
* diabetes, pregnancy, history of keloidal scarring; or patients with severe systemic illness or malignancy
* patients on anticoagulant therapy or aspirin or have a coagulation issue,
* patients with hemoglobin less than 10g\dl or platelet less than 105 micron\l
* any previous procedures for acne scar within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-10-20 (Actual)

PRIMARY OUTCOMES:
Change in Scar Appearance | Scar Appearance will be assessed at: T1; one day (wihtin 24 hours) before the application of the intervention(s); and T2: after three months of applying the intervention(s).

SECONDARY OUTCOMES:
Patients' Satisfaction | This is going to be assessed six months following the application of the intervention and the active comparator
  The assessment will be based on a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Faiez Al-Deghlaoui, MD MSc PhD, Study Director — Associate Professor of Dermatology and Veneology, Medical School, University of Damascus
Locations (1):
- Department of Dermatology and Venereology, Damascus, Syrian Arab Republic, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Layton AM, Henderson CA, Cunliffe WJ. A clinical evaluation of acne scarring and its incidence. Clin Exp Dermatol. 1994 Jul;19(4):303-8. doi: 10.1111/j.1365-2230.1994.tb01200.x. PMID 7955470
- [Background] Cunliffe WJ, Gould DJ. Prevalence of facial acne vulgaris in late adolescence and in adults. Br Med J. 1979 Apr 28;1(6171):1109-10. doi: 10.1136/bmj.1.6171.1109. PMID 156054
- [Background] Goulden V, Stables GI, Cunliffe WJ. Prevalence of facial acne in adults. J Am Acad Dermatol. 1999 Oct;41(4):577-80. PMID 10495379
- [Background] Sunitha Raja V, Munirathnam Naidu E. Platelet-rich fibrin: evolution of a second-generation platelet concentrate. Indian J Dent Res. 2008 Jan-Mar;19(1):42-6. doi: 10.4103/0970-9290.38931. PMID 18245923